CLINICAL TRIAL: NCT02449733
Title: Comprehensive HIV Prevention Package for MSM in Port Elizabeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Patrick S Sullivan, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB00079727
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: HIV
Keywords: voluntary counseling and testing (VCT); couples voluntary counseling and testing (CVCT); pre-exposure prophylaxis (PrEP); homosexuality; male; South Africa
MeSH Terms: conditions — Homosexuality | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; HIV Testing; Post-Exposure Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV+ subjects (Experimental): Men who test positive for HIV will receive a comprehensive package of HIV prevention services, including condom choices, condom-compatible lubricant choices, risk-reduction counseling, couples HIV counseling and testing, and linkage to care
  Interventions: Behavioral: Condom choices; Behavioral: Condom-compatible lubricant choices; Behavioral: Couples HIV counseling and testing (CVCT); Other: Linkage to care; Behavioral: Risk-reduction counseling
- HIV- subjects (Experimental): Men who test negative for HIV will receive a comprehensive package of HIV prevention services, including condom choices, condom-compatible lubricant choices, enhanced HIV testing options, risk-reduction counseling, couples HIV counseling and testing, linkage to care, and screening for and offering of pre-exposure prophylaxis (PrEP) and post-exposure prophylaxis (PEP).
  If men test positive for HIV during the study, they will be transitioned into the HIV+ subjects arm.
  Interventions: Behavioral: Condom choices; Behavioral: Condom-compatible lubricant choices; Behavioral: Couples HIV counseling and testing (CVCT); Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF); Other: HIV Testing; Other: Linkage to care; Procedure: Post-exposure prophylaxis (PEP); Behavioral: Risk-reduction counseling

INTERVENTIONS:
Behavioral: Condom choices — Men will receive the condom package that includes an assortment of styles, sizes, features and colors at their baseline visit, and will be able to get more condoms for free at any time after that visit by coming to a study clinic during clinic hours, or during a scheduled study visit.
Behavioral: Condom-compatible lubricant choices — Men will receive condom-compatible lubricant that will include different types of lubricant (e.g., silicone-based) and different packaging (individual sachets or flat, discreet packages) at their baseline study visit, and participants will be able to access enhanced condom-compatible lubricant at any time after that visit by coming to a study clinic during clinic hours, or during a scheduled study visit.
Behavioral: Couples HIV counseling and testing (CVCT) — Participants will be invited to schedule couples voluntary HIV counseling and testing (CVCT) appointments with a clinic counselor at any point after they complete their baseline study visit.
Drug: Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) — FTC/TDF is a once daily oral tablet taken with or without food. The tablet includes 200 mg of emtricitabine (FTC) and 300 mg of tenofovir disoproxil fumarate (TDF).
  For men who meet eligibility criteria, Pre-exposure prophylaxis (PrEP) with Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF) will be made available beginning one month into the study. Men who express interest and meet eligibility criteria at their baseline visit can initiate PrEP at 1 month if they test negative for HIV. For men with extenuating circumstances, whose risk profile changes, of those who become more comfortable with the PrEP intervention through enrollment in the study, PrEP will be available to initiate at the 4 month visit.
  Other Names: Truvada
  Arms: HIV- subjects
Other: HIV Testing — Rapid HIV testing at multiple time points
  Arms: HIV- subjects
Other: Linkage to care — Men will be linked to needed services including HIV care and treatment for positives identified at baseline or during the study, including antiretroviral medications, and mental health services. At the end of their baseline visit, participants will receive service referral handouts for HIV care and treatment, mental health services, and other resources, as appropriate. Men who test positive for sexually transmitted infections (STIs )will be treated at the clinic site.
Procedure: Post-exposure prophylaxis (PEP) — Two to three antiretroviral medicines as soon as possible (recommended is emtricitabine/tenofovir disoproxil fumarate plus either raltegravir or dolutegravir), but no more than 72 hours (3 days) after one may have been exposed to HIV, to try to reduce the chance of becoming HIV-positive. They must be taken for 28 days.
  Arms: HIV- subjects
Behavioral: Risk-reduction counseling — Risk-reduction counseling will be provided to all men at baseline and additionally at 3, 6, and 12 month visits, with an additional counseling session for men on PrEP at their initiation visit (either month 1 or 4), their 1-month follow-up visit (either month 2 or 5) and at their 9 month visit. Risk reduction counseling will be client-centered counseling, according to CDC's Fundamentals of HIV Prevention Counseling protocol.

SUMMARY:
The purpose of this study is to evaluate the acceptability and uptake of a combination package of biomedical, behavioral and community-level HIV prevention interventions and services for men who have sex with men (MSM) in South Africa.

DETAILED DESCRIPTION:
The objective of the Sibanye Health Project is to develop and evaluate a combination package of biomedical, behavioral and community-level HIV prevention interventions and services for men who have sex with men (MSM) in Africa. Experience implementing the prevention interventions and preliminary data collected regarding the acceptability of the HIV prevention package will be used to develop a proposal to design a larger efficacy trial to test the combination HIV prevention package for MSM.

ELIGIBILITY:
Inclusion Criteria:

* Male sex at birth
* Anal sex with another man in the past 12 months
* 18 years of age or older
* Resident of the study city, Port Elizabeth
* Able to complete study instruments, with or without assistance, in English, Xhosa or Afrikaans
* Willing to provide contact information
* Has a phone

Exclusion Criteria:

* Not male sex at birth
* No self-reported anal sex with a man in the past 12 months
* Less than 18 years of age
* Not a resident of the study city
* Plans to move from the study city within the year after enrollment
* Not able to complete study instructions, with or without assistance, in English, Xhosa or Afrikaans
* Not willing to provide contact information
* Does not have a phone

Additional Inclusion and Exclusion Criteria for participants on PrEP:

PrEP Inclusion Criteria:

* Identified as high-risk for HIV by the provider by meeting one or more of the criteria below:
* Have multiple partners
* Engage in transactional sex, including sex workers
* Use or abuse drugs
* Drink alcohol heavily
* Had more than 1 episode of a STI in the last year
* Is the HIV-negative partner in a discordant relationship, especially if the HIV-positive partner is not on antiretroviral therapy (ART)
* Is in a non-monogamous concordant relationship with a HIV-negative partner
* Is unable or unwilling to achieve consistent use of male condoms
* No contra-indications to Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF)
* Calculated creatinine clearance of at least 60 mL/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2 x upper limit of normal (ULN)
* Hepatitis B surface antigen (HBsAg) negative
* Motivated to follow PrEP prescribing guidelines
* Willing to adhere to daily oral dosing
* Willing to attend PrEP maintenance visits every 3 months

PrEP Exclusion Criteria:

* HIV positive
* Signs or symptoms suggestive of acute HIV infection
* Have baseline creatinine clearance <60 ml/min
* Are unwilling to follow PrEP prescribing guidelines
* Are unwilling to attend PrEP maintenance visits every 3 months
* Are known to have hypertensives or diabetes
* Are hepatitis B susceptible (test HBsAg and HBsAb negative) and refuse to take a hepatitis B vaccine series
* Any contraindication to taking FTC/TDF
* Proteinuria 2+ or greater at screening
* Glucosuria 2+ or greater at screening
* Use of antiretroviral (ARV) therapy (e.g., for PEP or PrEP) in the 90 days prior to study entry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Retention in the cohort | 12 months
  Will assess the ability of the study to retain participants for full study period. This will be measured by the proportion of enrolled participants who attend all subsequent study visits through the 12-month visit.
Use of PrEP | 6 months
  Will assess uptake of PrEP by study participants. This will be measured as the proportion of enrolled participants eligible for PrEP at the 3 and 6-month study visits who choose to initiate PrEP at those visits.
Incident HIV infection | 12 months
  This will be measured as the number of seroconversions during follow-up among those who are HIV-uninfected at baseline.

SECONDARY OUTCOMES:
Condom use | 3 months
  Measured as the proportion of anal intercourse that is protected by condoms in the prior 3 months as self-reported reported in the questionnaire at each study visit.
Lubricant use | 3 months
  Measured as the proportion of condom-protected anal intercourse in the prior for 3 months for which condom-compatible lubricant is used as self-reported in the questionnaire at each study visit.
VCT and CVCT uptake | 12 months
  Measured as the number of times participants report HIV testing in the study period as part of the study visits and outside study visits compared to the number of time participants reported HIV testing in the year prior at baseline.
Serodiscordant unprotected anal intercourse (UAI) | 3 months
  Measured as self-reported UAI in the last 3 months with a partner of positive or unknown HIV status as self-reported in the questionnaire at each study visit, pre- and post-intervention.
Acceptability of PEP | 12 months
  Measured as the proportion of men who report an eligible exposure who accept and initiate PEP.
MSM-specific provider training | 12 months
  Measured as the proportion of providers who are offered training who accept the training.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S Sulivan, DVM, PhD, Principal Investigator — Rollins School of Public Health; A.D. McNaghten, PhD, MHSA, Principal Investigator — Rollins School of Public Health; Stefan Baral, MD, MPH, CCFP, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Nancy Phaswanamafuya, PhD, Principal Investigator — Human Sciences Research Council
Locations (1):
- Human Sciences Research Council, Port Elizabeth, South Africa